CLINICAL TRIAL: NCT02117687
Title: A Safety and Efficacy Study of OPTIVE FUSION™ With VISMED® Multi for the Management of Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAF-AGN-OPH-DE-016
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPTIVE FUSION™ (Active Comparator): 1-2 drops OPTIVE FUSION™ (carboxymethylcellulose 0.5%/glycerin 0.9%) in each eye as needed at least 2 times and no more than 6 times daily, for 3 months.
  Interventions: Drug: carboxymethylcellulose 0.5%/glycerin 0.9%
- VISMED® Multi (Active Comparator): 1-2 drops VISMED® Multi (sodium hyaluronate 0.18%) in each eye as needed at least 2 times and no more than 6 times daily, for 3 months.
  Interventions: Drug: sodium hyaluronate 0.18%

INTERVENTIONS:
Drug: carboxymethylcellulose 0.5%/glycerin 0.9% — 1-2 drops OPTIVE FUSION™ (carboxymethylcellulose 0.5%/glycerin 0.9%) in each eye as needed at least 2 times and no more than 6 times daily, for 3 months.
  Other Names: OPTIVE FUSION™
  Arms: OPTIVE FUSION™
Drug: sodium hyaluronate 0.18% — 1-2 drops VISMED® Multi (sodium hyaluronate 0.18%) in each eye as needed at least 2 times and no more than 6 times daily, for 3 months.
  Other Names: VISMED® Multi
  Arms: VISMED® Multi

SUMMARY:
This study will evaluate the safety and efficacy of OPTIVE FUSION™ compared to VISMED® Multi for the management of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Use of artificial tears for dry eye in both eyes for at least 3 months
* Use of preservative-free artificial tears at least twice daily for 2 weeks;

Exclusion Criteria:

* Cataract, laser-assisted in situ keratomileusis (LASIK), photorefractive keratectomy (PRK) surgery in the last 12 months
* Use of punctal plugs or contact lenses in the last month
* Active ocular allergy within last 2 years
* Best corrected visual acuity (BCVA) less than 20/200 in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2015-01-27 (Actual); Study Completion 2015-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Paris, France
- London, United Kingdom

REFERENCES:
- [Background] Labetoulle M, Chiambaretta F, Shirlaw A, Leaback R, Baudouin C. Osmoprotectants, carboxymethylcellulose and hyaluronic acid multi-ingredient eye drop: a randomised controlled trial in moderate to severe dry eye. Eye (Lond). 2017 Oct;31(10):1409-1416. doi: 10.1038/eye.2017.73. Epub 2017 Apr 28. PMID 28452989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Started | 40 | 40
Completed | 39 | 36
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Other Reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPTIVE FUSION™ | VISMED® Multi | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Customized [Number; unit: Participants]
  <65 years | 17 | 25 | 42
  ≥65 years | 23 | 15 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Global Ocular Staining Score in the Study Eye
Description: Global ocular staining of the study eye was graded from 0 to 15 and was the sum of corneal fluorescein staining severity, nasal conjunctiva lissamine green staining severity, and temporal conjunctiva lissamine green staining severity. Staining of the cornea followed ocular administration of fluorescein dye and was graded on a 6-point scale (0=no staining to 5=diffuse staining). Staining of the conjunctiva followed ocular administration of lissamine green dye and was graded on a 6-point scale (0=no staining to 5=diffuse staining). Conjunctival staining was evaluated in two zones, nasal and temporal.
Time Frame: Baseline, Day 35
Population: Per Protocol: all randomized subjects who received at least one dose of the study product, had at least one follow-up visit, and who did not adhere to a pre-defined list of protocol violation criteria
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Baseline | 5.2 (1.11) | 5.2 (1.21)
  Change from Baseline at Day 35 | -1.5 (1.54) | -1.6 (1.54)

2. Secondary Outcome: Change From Baseline in Global Ocular Staining Score in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Baseline | 5.2 (1.11) | 5.2 (1.21)
  Change from Baseline at Day 35 | -2.5 (2.23) | -2.4 (2.24)

3. Secondary Outcome: Change From Baseline in Ocular Surface Disease Index© (OSDI) Score
Description: The OSDI is a 12-question survey for patients to document their dry eye disease symptoms on a 5-point scale (0=none of the time and 4=all of the time). Higher scores represent greater disability. Scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability and 100=complete disability). A negative number change from baseline represents an improvement and a positive number change from baseline represents a worsening.
Time Frame: Baseline, Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Baseline | 45.5 (22.02) | 44.4 (17.60)
  Change from Baseline at Day 35 | -10.3 (13.51) | -12.9 (13.13)

4. Secondary Outcome: Change From Baseline in the Schirmer Test in the Study Eye
Description: The Schirmer's Test measures the rate of secretion of tears produced by the study eye over 5 minutes. The results indicate the presence of dry eye (Normal = greater than or equal to 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye. A positive number change from baseline indicates an increase in tears (improvement) and a negative number change from baseline indicates a decrease in tears (worsening).
Time Frame: Baseline, Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters (mm)/5 Minutes
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Millimeters (mm)/5 Minutes
  Baseline | 11.1 (10.22) | 8.7 (7.29)
  Change from Baseline at Day 35 | 0.1 (7.74) | 1.0 (5.44)

5. Secondary Outcome: Subject Assessment of Dry Eye Symptoms on a 5-Point Scale
Description: Subjects assess dry eye symptoms on a 5-point scale (none, mild, moderate, severe, very severe).
Time Frame: Baseline, Day 35, Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Subjects
  Baseline Stinging/Burning - None (N=32,28) | 0 | 1
  Baseline Stinging/Burning - Mild (N=32,28) | 7 | 4
  Baseline Stinging/Burning - Moderate (N=32,28) | 17 | 13
  Baseline Stinging/Burning - Severe (N=32,28) | 7 | 9
  Baseline Stinging/Burning - Very Severe (N=32,28) | 1 | 1
  Day 35 Stinging/Burning - None | 5 | 2
  Day 35 Stinging/Burning - Mild | 12 | 8
  Day 35 Stinging/Burning - Moderate | 17 | 17
  Day 35 Stinging/Burning - Severe | 1 | 3
  Day 35 Stinging/Burning - Very Severe | 0 | 1
  Month 3 Stinging/Burning - None | 5 | 6
  Month 3 Stinging/Burning - Mild | 14 | 5
  Month 3 Stinging/Burning - Moderate | 15 | 13
  Month 3 Stinging/Burning - Severe | 1 | 6
  Month 3 Stinging/Burning - Very Severe | 0 | 1
  Baseline Itching - None (N=32,28) | 6 | 5
  Baseline Itching - Mild (N=32,28) | 8 | 7
  Baseline Itching - Moderate (N=32,28) | 12 | 1
  Baseline Itching - Severe (N=32,28) | 6 | 3
  Baseline Itching - Very Severe (N=32,28) | 0 | 2
  Day 35 Itching- None | 10 | 8
  Day 35 Itching- Mild | 8 | 7
  Day 35 Itching- Moderate | 15 | 13
  Day 35 Itching- Severe | 2 | 2
  Day 35 Itching- Very Severe | 0 | 1
  Month 3 Itching- None | 10 | 10
  Month 3 Itching- Mild | 12 | 8
  Month 3 Itching- Moderate | 11 | 9
  Month 3 Itching- Severe | 2 | 3
  Month 3 Itching- Very Severe | 0 | 1
  Baseline Sandiness/Grittiness - None (N=32,28) | 2 | 1
  Baseline Sandiness/Grittiness - Mild (N=32,28) | 6 | 5
  Baseline Sandiness/Grittiness - Moderate (N=32,28) | 19 | 12
  Baseline Sandiness/Grittiness - Severe (N=32,28) | 5 | 8
  Bsln Sandiness/Grittiness-Very Severe (N=32,28) | 0 | 2
  Day 35 Sandiness/Grittiness - None | 7 | 4
  Day 35 Sandiness/Grittiness - Mild | 13 | 8
  Day 35 Sandiness/Grittiness - Moderate | 14 | 13
  Day 35 Sandiness/Grittiness - Severe | 1 | 4
  Day 35 Sandiness/Grittiness - Very Severe | 0 | 2
  Month 3 Sandiness/Grittiness - None | 7 | 8
  Month 3 Sandiness/Grittiness - Mild | 17 | 4
  Month 3 Sandiness/Grittiness - Moderate | 9 | 15
  Month 3 Sandiness/Grittiness - Severe | 2 | 3
  Month 3 Sandiness/Grittiness - Very Severe | 0 | 1
  Baseline Blurred Vision - None (N=32,28) | 11 | 10
  Baseline Blurred Vision - Mild (N=32,28) | 8 | 7
  Baseline Blurred Vision - Moderate (N=32,28) | 10 | 7
  Baseline Blurred Vision - Severe (N=32,28) | 3 | 3
  Baseline Blurred Vision - Very Severe (N=32,28) | 0 | 1
  Day 35 Blurred Vision - None | 16 | 13
  Day 35 Blurred Vision - Mild | 10 | 9
  Day 35 Blurred Vision - Moderate | 8 | 7
  Day 35 Blurred Vision - Severe | 1 | 1
  Day 35 Blurred Vision - Very Severe | 0 | 1
  Month 3 Blurred Vision - None | 20 | 14
  Month 3 Blurred Vision - Mild | 7 | 9
  Month 3 Blurred Vision - Moderate | 6 | 5
  Month 3 Blurred Vision - Severe | 1 | 1
  Month 3 Blurred Vision - Very Severe | 1 | 2
  Baseline Dryness - None (N=32,28) | 1 | 1
  Baseline Dryness - Mild (N=32,28) | 2 | 2
  Baseline Dryness - Moderate (N=32,28) | 13 | 10
  Baseline Dryness - Severe (N=32,28) | 13 | 12
  Baseline Dryness - Very Severe (N=32,28) | 3 | 3
  Day 35 Dryness - None | 4 | 3
  Day 35 Dryness - Mild | 8 | 5
  Day 35 Dryness - Moderate | 16 | 14
  Day 35 Dryness - Severe | 7 | 7
  Day 35 Dryness - Very Severe | 0 | 2
  Month 3 Dryness - None | 2 | 3
  Month 3 Dryness - Mild | 12 | 5
  Month 3 Dryness - Moderate | 17 | 14
  Month 3 Dryness - Severe | 4 | 6
  Month 3 Dryness - Very Severe | 0 | 3
  Baseline Light Sensitivity - None (N=32,28) | 1 | 2
  Baseline Light Sensitivity - Mild (N=32,28) | 4 | 8
  Baseline Light Sensitivity - Moderate (N=32,28) | 14 | 6
  Baseline Light Sensitivity - Severe (N=32,28) | 9 | 7
  Baseline Light Sensitivity - Very Severe (N=32,28) | 4 | 5
  Day 35 Light Sensitivity - None | 5 | 2
  Month 3 Light Sensitivity - Severe | 5 | 8
  Month 3 Light Sensitivity - Very Severe | 1 | 3
  Day 35 Light Sensitivity - Mild | 6 | 7
  Day 35 Light Sensitivity - Moderate | 18 | 11
  Day 35 Light Sensitivity - Severe | 5 | 7
  Day 35 Light Sensitivity - Very Severe | 1 | 4
  Month 3 Light Sensitivity - None | 5 | 2
  Month 3 Light Sensitivity - Mild | 16 | 10
  Month 3 Light Sensitivity - Moderate | 8 | 8
  Baseline Painful or Sore - None (N=31,28) | 0 | 1
  Baseline Painful or Sore - Mild (N=31,28) | 12 | 8
  Baseline Painful or Sore - Moderate (N=31,28) | 15 | 13
  Baseline Painful or Sore - Severe (N=31,28) | 4 | 4
  Baseline Painful or Sore - Very Severe (N=31,28) | 0 | 2
  Day 35 Painful or Sore - None | 5 | 5
  Day 35 Painful or Sore - Mild | 20 | 9
  Day 35 Painful or Sore - Moderate | 9 | 13
  Day 35 Painful or Sore - Severe | 1 | 2
  Day 35 Painful or Sore - Very Severe | 0 | 2
  Month 3 Painful or Sore - None | 5 | 9
  Month 3 Painful or Sore - Mild | 17 | 3
  Month 3 Painful or Sore - Moderate | 10 | 16
  Month 3 Painful or Sore - Severe | 2 | 2
  Month 3 Painful or Sore - Very Severe (N=34,31) | 0 | 1
  Baseline Other - None (N=3,1) | 0 | 0
  Baseline Other - Mild (N=3,1) | 0 | 0
  Baseline Other - Moderate (N=3,1) | 1 | 0
  Baseline Other - Severe (N=3,1) | 0 | 0
  Baseline Other - Very Severe (N=3,1) | 0 | 1
  Day 35 Other - None (N=1,3) | 0 | 0
  Day 35 Other - Mild (N=1,3) | 0 | 0
  Day 35 Other - Moderate (N=1,3) | 1 | 1
  Day 35 Other - Severe (N=1,3) | 0 | 1
  Day 35 Other - Very Severe (N=1,3) | 0 | 1
  Month 3 Other - None (N=1,3) | 0 | 1
  Month 3 Other - Mild (N=1,3) | 0 | 0
  Month 3 Other - Moderate (N=1,3) | 1 | 0
  Month 3 Other - Severe (N=1,3) | 0 | 1
  Month 3 Other - Very Severe (N=1,3) | 0 | 1

6. Secondary Outcome: Subject Global Assessment of Treatment Efficacy on a 5-Point Scale
Description: Subjects assess global treatment efficacy compared to baseline on a 5-point scale (much worse, worse, about the same, improved, much improved).
Time Frame: Baseline, Day 35, Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Subjects
  Day 35 - Much Worse | 0 | 0
  Day 35 - Worse | 0 | 3
  Day 35 - About the Same | 12 | 11
  Day 35 - Improved | 21 | 14
  Day 35 - Much Improved | 2 | 3
  Month 3 - Much Worse | 0 | 1
  Month 3 - Worse | 0 | 3
  Month 3 - About the Same | 11 | 10
  Month 3 - Improved | 19 | 13
  Month 3 - Much Improved | 5 | 4

7. Secondary Outcome: Subject Assessment of Treatment Acceptability on a 5-Point Scale
Description: Subjects assess treatment acceptability (likability and comfort) on a 5-point scale (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree).
Time Frame: Day 35
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Subjects
  Liked - Strongly Agree (N=35,30) | 14 | 8
  Liked - Agree (N=35,30) | 12 | 10
  Liked - Neither Agree nor Disagree (N=35,30) | 6 | 9
  Liked - Disagree (N=35,30) | 2 | 2
  Liked - Strongly Disagree (N=35,30) | 1 | 1
  Comfortable - Strongly Agree | 9 | 9
  Comfortable - Agree | 16 | 13
  Comfortable - Neither Agree nor Disagree | 7 | 6
  Comfortable - Disagree | 2 | 2
  Comfortable - Strongly Disagree | 1 | 1

8. Secondary Outcome: Investigator Global Assessment of Treatment Efficacy on a 4-Point Scale
Description: Investigators assess global treatment efficacy on a 4-point scale (very satisfactory, satisfactory, poor, very poor).
Time Frame: Day 35, Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Subjects
  Day 35 - Very Satisfactory | 13 | 8
  Day 35 - Satisfactory | 17 | 19
  Day 35 - Poor | 5 | 4
  Day 35 - Very Poor | 0 | 0
  Month 3 - Very Satisfactory | 15 | 10
  Month 3 - Satisfactory | 15 | 11
  Month 3 - Poor | 5 | 9
  Month 3 - Very Poor | 0 | 1

9. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT) in the Study Eye
Description: TBUT is the time required for dry spots to appear on the surface of the eye after blinking in the worse eye. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement) and a negative number change from baseline indicates a decrease in TBUT (worsening).
Time Frame: Baseline, Day 35
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Seconds
  Baseline | 5.52 (2.575) | 5.75 (3.146)
  Change from Baseline at Day 35 | 0.6 (1.66) | 0.7 (2.00)

10. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire Score
Description: The Work Productivity and Activity questionnaire assesses the effect of dry eye on the ability of subjects to work and perform regular activities on a scale from 0 to 10 during the past 7 days (0=dry eye had no effect on my work/daily activities to 10=dry eye completely prevented me from working/doing my daily activities). Since not all subjects were in full time employment during the study, not all items of the questionnaire were applicable to all subjects at each visit. Outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Day 35, Month 3
Population: Per Protocol: all randomized subjects who received at least one dose of the study product, had at least one follow-up visit, who did not adhere to a pre-defined list of protocol violation criteria, and who had data for this data point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Baseline - Work Productivity (N=11,13) | 3.09 (1.921) | 3.46 (3.382)
  Baseline - Activity Impairment | 3.91 (2.035) | 4.35 (2.550)
  Day 35 - Work Productivity (N=11,9) | 2.55 (1.809) | 2.33 (1.936)
  Day 35 - Activity Impairment (N=34,31) | 3.09 (2.065) | 3.52 (2.393)
  Month 3 - Work Productivity (N=11,10) | 1.82 (0.982) | 2.40 (2.066)
  Month 3 - Activity Impairment | 2.14 (1.630) | 2.77 (2.232)

11. Secondary Outcome: Change From Baseline in Corneal Staining in the Study Eye
Description: The cornea is the transparent front part of the eye which covers the iris and pupil. Staining of the cornea followed ocular administration of fluorescein dye and was graded on a 6-point scale (0=no staining to 5=diffuse staining). A negative number change from baseline represents a decrease in corneal staining (improvement) and a positive number change from baseline represents an increase in corneal staining (worsening).
Time Frame: Baseline, Day 35, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Baseline | 1.7 (0.68) | 1.9 (0.65)
  Change from Baseline at Day 35 | -0.4 (0.77) | -0.7 (0.83)
  Change from Baseline at Month 3 | -0.8 (0.84) | -0.9 (1.04)

12. Secondary Outcome: Change From Baseline in Conjunctival Staining in the Study Eye
Description: The conjunctiva is the clear membrane covering the white surface of the eye. Staining of the conjunctiva followed ocular administration of lissamine green dye and was graded on a 6-point scale (0=no staining to 5=diffuse staining) in the temporal and nasal locations. A negative number change from baseline represents a decrease in corneal staining (improvement) and a positive number change from baseline represents an increase in corneal staining (worsening).
Time Frame: Baseline, Day 35, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Scores on a Scale
  Baseline - Temporal | 1.7 (0.64) | 1.6 (0.81)
  Change from Baseline at Day 35 - Temporal | -0.5 (0.66) | -0.5 (0.81)
  Change from Baseline at Month 3 - Temporal | -0.8 (0.79) | -0.8 (0.92)
  Baseline - Nasal | 1.9 (0.66) | 1.7 (0.70)
  Change from Baseline at Day 35 - Nasal | -0.6 (0.65) | -0.5 (0.68)
  Change from Baseline at Month 3 - Nasal | -0.9 (0.97) | -0.7 (0.87)

13. Secondary Outcome: Conjunctival Hyperaemia in the Study Eye
Description: Macroscopic conjunctival hyperemia (eye redness) is graded in the study eye on a 5-point scale (none, trace, mild, moderate, severe).
Time Frame: Baseline, Day 35, Month 3
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Subjects
  Baseline - None | 8 | 8
  Baseline - Trace | 13 | 11
  Baseline - Mild | 13 | 10
  Baseline - Moderate | 1 | 2
  Baseline Severe | 0 | 0
  Day 35 - None | 17 | 12
  Day 35 - Trace | 9 | 10
  Day 35 - Mild | 9 | 8
  Day 35 - Moderate | 0 | 1
  Day 35 - Severe | 0 | 0
  Month 3 - None | 22 | 14
  Month 3 - Trace | 8 | 7
  Month 3 - Mild | 5 | 9
  Month 3 - Moderate | 0 | 1
  Month 3 - Severe | 0 | 0

14. Secondary Outcome: Study Product Use
Description: The number of times the study product is administered per day is recorded.
Time Frame: Day 8, Day 35, Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Times/Day
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Number analyzed (Participants) | 35 | 31
Number of Times/Day
  Day 8 | 3.63 (1.190) | 3.47 (0.900)
  Day 35 | 3.77 (1.285) | 3.39 (0.761)
  Month 3 | 3.71 (1.178) | 3.42 (0.958)

ADVERSE EVENTS:
Description: The Safety Population included all randomized subjects treated with at least one dose of study product. The Safety Population was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | OPTIVE FUSION™ | VISMED® Multi
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/40
Other Adverse Events (participants affected / at risk) | 4/40 | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPTIVE FUSION™ (N=40) | VISMED® Multi (N=40)
Pericarditis (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPTIVE FUSION™ (N=40) | VISMED® Multi (N=40)
Dry Eye (Eye disorders) | 0 | 2
Eye Discharge (Eye disorders) | 0 | 2
Eye Irritation (Eye disorders) | 2 | 2
Eye Pruritus (Eye disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.